CLINICAL TRIAL: NCT04179968
Title: The Role of 68Gallium PSMA-11 in Enhancing Diagnosis of Primary and Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana Mathews (Other)
Responsible Party: Sponsor-Investigator, Dana Mathews, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2019-1198
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic
Keywords: PET/CT; prostate cancer; Gallium-68; PSMA-11
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Unblinded, single arm imaging study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with suspected prostate cancer (Experimental): Patients with suspected prostate cancer who have at least one PI-RADS 5 lesion, or at least one PI-RADS 4 lesion and PSA ≥10 nanograms/milliliter (ng/mL), on standard of care mpMRI of the prostate, who are scheduled for biopsy or radical prostatectomy
  Interventions: Drug: 68Ga PSMA-11 injection; Procedure: Positron Emission Tomography/Computed Tomography

INTERVENTIONS:
Drug: 68Ga PSMA-11 injection — Injection of 68Ga PSMA-11
Procedure: Positron Emission Tomography/Computed Tomography — PET/CT scan after 68Ga PSMA-11 injection
  Other Names: PET/CT

SUMMARY:
To goal of this research is to assess the ability of Gallium-68 (68Ga) Prostate-Specific Membrane Antigen-11 (PSMA-11) positron emission tomography/computed tomography (PET/CT) to increase diagnostic accuracy in localizing primary and metastatic lesions in patients with suspected prostate cancer and elevated Prostate Imaging Reporting and Data System (PI-RADS) scores and Prostate-Specific Antigen (PSA).

DETAILED DESCRIPTION:
This study is designed to evaluate the added value of 68Ga PSMA-11 PET/CT for detection of additional primary prostate cancer lesions compared to multiparametric magnetic resonance imaging (mpMRI) in a group of patients with elevated PI-RADS scores and PSA. We propose that the addition of early dynamic 68Ga PSMA-11 PET/CT imaging to the more usual delayed imaging will enhance detection of primary lesions and additional lesions not detected on the mpMRI. In addition, the dynamic imaging will allow us to evaluate the kinetics of uptake in the prostate gland. It is possible that even in the absence of focal uptake, hyperemia of the gland could indicate the presence of an occult primary.

A second purpose of this research is to examine the value of 68Ga PSMA-11 PET/CT in this same group of patients in detecting metastatic disease at initial staging in comparison with current standard of care imaging such as computed tomography (CT) and magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected prostate cancer (e.g., abnormal digital rectal exam, elevated and/or rising PSA) as determined by referring physician
* Patients must have had a diagnostic, standard of care mpMRI of the prostate with at least one lesion with a PI-RADS v2.1 score ≥ 4
* In men with PI-RADS v2.1 score 4, PSA should be ≥ 10 ng/mL. In men with at least one PI-RADS v2.1 score 5 lesion, there is no restriction on PSA level.
* Patients must be scheduled for biopsy or radical prostatectomy
* Patients should not have had any type of curative or palliative therapy for prostate cancer before enrolling in the study
* Patients must be medically stable as judged by the patient's physician
* Patients must be able to lie still for a total of 60 minutes for the PET/CT scans
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who have had a prior prostatectomy or radiotherapy for prostate cancer cannot participate in the study
* Patients who have had a prior biopsy for prostate cancer cannot participate in the study
* Patients who have been treated for cancers other than skin cancers
* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study
* Patients may not weigh more than the maximum weight limit for the PET/CT scanner table (>200 kilograms or 440 pounds)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 68Ga PSMA-11 or other agents used in the study such as gadolinium-based intravenous contrast agent used during the mpMRI
* Prior transurethral resection of the prostate (TURP)/benign prostatic hyperplasia (BPH) procedures, including steam/laser therapies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orhan K Oz, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parrott D, Yuan Q, Pinho D, Xi Y, Costa DN, De Leon AD, Dakanali M, Sun X, Oz OK, Bowen S, Rofsky NM, Mathews D, Pedrosa I. Characterization of suspicious prostate lesions at multiparametric MRI with dynamic 68 Ga-Gozetotide PET/CT. EJNMMI Rep. 2025 Oct 13;9(1):35. doi: 10.1186/s41824-025-00268-2. PMID 41077599

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Suspected Prostate Cancer: Patients with suspected prostate cancer who have at least one Prostate Imaging Reporting & Data System (PI-RADS) 5 lesion, or at least one PI-RADS 4 lesion and prostate-specific antigen (PSA) ≥10 nanograms/milliliter (ng/mL), on standard of care multiparametric (mpMRI) of the prostate, who are scheduled for biopsy or radical prostatectomy
  68Gallium (68Ga) prostate-specific membrane antigen-11 (PSMA-11) injection: Injection of 68Ga PSMA-11
  Positron Emission Tomography (PET)/Computed Tomography (CT): PET/CT scan after 68Ga PSMA-11 injection
Period: Overall Study
Arm/Group | Patients With Suspected Prostate Cancer
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Suspected Prostate Cancer
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.85 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Primary Prostate Lesions Detected on Early Dynamic 68Ga-PSMA-11 PET/CT Imaging
Description: Number of primary prostate lesions will be detected using early dynamic 68Ga-PSMA-11 PET/CT imaging. PSMA is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protein.
Time Frame: During PET/CT imaging, up to 2 hours
Population: All patients who received a 68Ga-PSMA-11 injection for diagnosis of primary prostate cancer with PET/CT imaging.
Measure: Number; unit: lesions
Arm/Group | Patients With Suspected Prostate Cancer
Number analyzed (Participants) | 19
lesions | 24

2. Primary Outcome: Number of Primary Prostate Lesions Detected by mpMRI
Description: Number of primary prostate lesions will be detected by using mpMRI.
Time Frame: During mpMRI, up to 2 hours
Population: All patients who received a 68Ga-PSMA-11 injection for diagnosis of primary prostate cancer with PET/CT imaging.
Measure: Number; unit: lesions
Arm/Group | Patients With Suspected Prostate Cancer
Number analyzed (Participants) | 19
lesions | 37

3. Secondary Outcome: Number of Sites of Metastatic Prostate Lesions Detected on 68Ga-PSMA-11 PET/CT
Description: Number of sites of metastatic prostate lesions will be detected using 68Ga-PSMA-11 PET/CT. PSMA is a protein expressed on prostate cancer cells that can be imaged using small molecules that target this protein.
Time Frame: During PET/CT imaging, up to 2 hours
Population: 19 patients completed 68Ga-PSMA-11 PET/CT imaging as part of the study.
Measure: Number; unit: sites
Arm/Group | Patients With Suspected Prostate Cancer
Number analyzed (Participants) | 19
sites | 7

4. Secondary Outcome: Number of Sites of Metastatic Prostate Lesions Detected by Current Standard of Care Imaging (CT/MRI)
Description: Patients with metastatic prostate lesions were imaged using current standard of care imaging (CT/MRI).
Time Frame: During CT/MRI imaging, up to 2 hours
Population: All patients who received a 68Ga-PSMA-11 injection for diagnosis of primary prostate cancer with PET/CT imaging
Measure: Number; unit: sites
Arm/Group | Patients With Suspected Prostate Cancer
Number analyzed (Participants) | 19
sites | 5

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events after injection of the investigational agent and were contacted 24 hours after completion of PET/CT imaging to assess any potentially related adverse events.
Arm/Group | Patients With Suspected Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Suspected Prostate Cancer (N=20)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea without emesis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT04179968/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04179968/ICF_001.pdf